CLINICAL TRIAL: NCT01718080
Title: The Role of Puberty and Insulin Resistance in the Development of Hyperglucagonemia
Brief Title: The Effects of Puberty and Weight on Sugar Metabolism in Children
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Luisa M. Rodriguez, The Role of Puberty and Insulin Resistance in the Development of Hyperglucagonemia, Baylor College of Medicine
Other Study IDs: H-29652; NIH 1K126K63691 (Other: NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Overweight; Leanness; Adolescent
Keywords: Obese, Lean, Pubertal, Prepubertal, Glucose, Adolescents, Type 2 Diabetes
MeSH Terms: conditions — Overweight; Thinness; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Healthy lean children before puberty
- Group B: Otherwise healthy overweight children before puberty
- Group C: Healthy lean adolescents in mid to late puberty
- Group D: Otherwise healthy overweight adolescents in mid to late puberty

SUMMARY:
Our goal is to investigate how hormones that control blood sugar, hunger, and stomach emptying change with puberty and being overweight. These substances change with a meal.

* For this, we need to compare lean and overweight children.
* We need to study them before and during puberty.
* All children in the study will be tested before and after a liquid meal.

ELIGIBILITY:
Inclusion Criteria:

All groups:

Healthy lean and otherwise healthy overweight children and adolescents between the ages of 8 and 17.

Exclusion Criteria:

Same for all groups

The subjects will be excluded if they have:

* a history of chronic disease
* allergy to acetaminophen
* evidence or history of chemical abuse
* abnormal lab values
* pregnancy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prepubertal and pubertal subjects.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overweight and Lean Children Sugar Metabolism Before and During Puberty | 4 hours
  Too much weight gain can cause changes in the substances that control blood sugar and hunger in the body. Scientists need to compare these substances in lean and overweight children before and during puberty. These substances can be measured before and after a meal in the blood and in the urine. The way your stomach moves food can change your sugar levels. We want to understand how diabetes develops by studying these things. This can help find better ways to prevent and treat diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa M. Rodriguez, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No